CLINICAL TRIAL: NCT05141318
Title: Family Reported Outcomes in the Estimation of Societal Value of Advanced Therapy Medicinal Products (ATMPs)
Brief Title: Evaluation of FROM-16 in ATMP Patients & Families
Status: Completed | Type: Observational
Sponsor: Swansea University (Other)
Collaborators: Cardiff University (Other); University of Hertfordshire (Other); Cardiff and Vale University Health Board (Other Government); University Hospital Birmingham NHS Foundation Trust (Other); University Hospitals, Leicester (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: WBS-ITT-43652
Record Dates: First submitted 2021-11-22; First posted 2021-12-02 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2021-11

CONDITIONS: Family Members; Cancer
Keywords: Family members; ATMPs; Family reported outcome measures; Value-based healthcare; Severe disease; Familial impact; Societal value; Advanced Therapy Medicinal Products
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FROM-16 Questionnaire — A 16-item questionnaire to provide information about the impact of a patient's disease/condition the participants (family member of patient) quality of life
Other: Semi-structured two-part interview — A telephone/video interview to provide additional context to the FROM-16 responses

SUMMARY:
Poor health, and its treatment, has impact beyond the healthcare system into wider society. A person's productivity, taxable earnings, benefit payments and community contribution may all be adversely affected by poor health. Family members living with or caring for a patient may suffer equally, or sometimes more than the patient themselves, but this familial burden has gone largely unrecognised by healthcare systems. The Family-Reported Outcome Measure (FROM-16) is the first generic questionnaire designed to measure the impact of any chronic disease on the quality of life of family members or partners of patients with a health condition. Advance Therapy Medicinal Products (ATMPs) are a novel & ground-breaking therapeutic approach for curative treatment of disease and/or injury where conventional treatments have been ineffective. Such disease/injury generally has an extremely high impact on the patient's quality of life, and also the quality of life of the patient's family, in particular those family members who take on the role of 'informal carer'. ATMPs usually have very high costs and this can limit their usage, especially in the context of low prevalence disease and publicly-funded healthcare systems, where healthcare providers may be reluctant to take on the cost burden of the ATMP therapy. As a result, there is a particular focus on the 'value' of ATMPs. An important component of value is 'Societal Value', where a treatment leads to societal contributions, and considering Societal Value may justify the high cost of ATMPs despite the relatively few patients cured. In this study, we will validate the FROM-16 for use as one measure of the Societal Value of very high cost, potentially curative treatments such as ATMPs.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patients of any age
* Ability to read English or Welsh (where age-appropriate).
* Capacity to give written informed consent, or assent for their family member to participate
* Attending ATMP treatment centre with a family member/carer.
* Being considered for, or have recently received, ATMP therapy for any diagnosed condition.

Family Members:

* Considered by the patient to be the person most affected by the patient's condition
* Adult family members aged 18 years or older.
* A family member or partner, living with or caring for, a patient who is being prepared to receive ATMP treatment or has recently received ATMP therapy for any diagnosed condition.
* Have capacity to give written informed consent and complete the interview and questionnaires.

Exclusion Criteria:

Patients:

* Adult patients: Lacking capacity, or unwilling to give written informed consent for their family member to participate.
* Gillick competent paediatric patients: unwilling to give written informed assent and/or consent for their family member to participate.
* Non-Gillick competent paediatric patients: patient's parent/guardian refuses to give consent or is unable to give consent on their behalf.
* Not being prepared for ATMP therapy, or is currently receiving ATMPs.

Family Members:

* Family members under 18 years of age.
* Not considered by the patient to be a family member or carer.
* Lacking capacity or willingness to give informed written consent to participate
* Having a severe handicap or disability that prevents the completion of interview and questionnaires.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Family members of patients, of any age, with diagnosed long-term diseases who are being prepared for ATMP therapy, or have completed an ATMP therapy, in ATMP provider centres primarily within the extended Midlands-Wales Advanced Therapy Treatment Centre (ATTC) network.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Validity of the FROM-16 to the ATMP population | November 2021 - March 2022
  Successful outcomes will be defined by this study demonstrating that the FROM-16 is a suitable tool for gathering FROMs from ATMP patient family members, through showing high reliability of the responses to the FROM-16, and showing that the FROM-16 is valid when applied to this population.
  Reliability, assessed by Cronbach's Alpha, should have scores in excess of 0.8, indicating high internal consistency.
  Validity will be assessed in three dimensions: Face, Construct and Content Validity. Face validity will be assessed by an experimenter independent to the data analytics and collection processes. Content validity will be assessed by thematic analysis of interview transcripts, and by assessing the intraclass correlation of themes. Construct validity will be assessed by measuring convergent and discriminatory validity by confirmatory factor analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hamish Laing, Principal Investigator — Swansea University
Locations (5):
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust1, Bristol
  - Cardiff & Vale University LHB, Cardiff
  - University Hospitals of Leicester NHS Trust, Leicester
  - Swansea University School of Management, Swansea

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers outside of the study team

REFERENCES:
- [Background] Golics CJ, Basra MK, Finlay AY, Salek S. The development and validation of the Family Reported Outcome Measure (FROM-16)(c) to assess the impact of disease on the partner or family member. Qual Life Res. 2014 Feb;23(1):317-26. doi: 10.1007/s11136-013-0457-y. PMID 23797564
- [Background] Golics CJ, Basra MK, Finlay AY, Salek S. The impact of disease on family members: a critical aspect of medical care. J R Soc Med. 2013 Oct;106(10):399-407. doi: 10.1177/0141076812472616. Epub 2013 May 10. PMID 23759884
- [Background] Golics CJ, Basra MK, Salek MS, Finlay AY. The impact of patients' chronic disease on family quality of life: an experience from 26 specialties. Int J Gen Med. 2013 Sep 18;6:787-98. doi: 10.2147/IJGM.S45156. eCollection 2013. PMID 24092994
- [Background] Goula A, Gkioka V, Michalopoulos E, Katsimpoulas M, Noutsias M, Sarri EF, Stavropoulos C, Kostakis A. Advanced Therapy Medicinal Products Challenges and Perspectives in Regenerative Medicine. J Clin Med Res. 2020 Dec;12(12):780-786. doi: 10.14740/jocmr3964. Epub 2020 Dec 18. PMID 33447311
- [Background] Chantarasap P, Johns NP, Pairojkul S, Sookprasert A, Wirasorn K, Cheawchanwattana A, Salek S, Subongkot S. Validation of the Thai version of the family reported outcome measure (FROM-16)(c) to assess the impact of disease on the partner or family members of patients with cancer. Health Qual Life Outcomes. 2019 Feb 8;17(1):32. doi: 10.1186/s12955-019-1091-3. PMID 30736795
- [Background] Basra MK, Sue-Ho R, Finlay AY. The Family Dermatology Life Quality Index: measuring the secondary impact of skin disease. Br J Dermatol. 2007 Mar;156(3):528-38. doi: 10.1111/j.1365-2133.2006.07617.x. PMID 17300244
- [Background] Brittain E, Muirhead N, Finlay AY, Vyas J. Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS): Major Impact on Lives of Both Patients and Family Members. Medicina (Kaunas). 2021 Jan 7;57(1):43. doi: 10.3390/medicina57010043. PMID 33430175
- See also: Description of Value-based healthcare — https://op.europa.eu/en/publication-detail/-/publication/beaebce1-ac29-11e9-9d01-01aa75ed71a1/language-en